CLINICAL TRIAL: NCT04967885
Title: Evaluation of an Ecological Momentary Intervention of Implementation Intentions Delivered by Text Message to Reduce Cigarette Smoking
Brief Title: Ecological Momentary Intervention of Implementation Intentions Delivered by Text Message to Reduce Cigarette Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 10836; 5P30DA029926 (NIH)
Record Dates: First submitted 2021-07-08; First posted 2021-07-20 (Actual); Results first posted 2023-03-27 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-03

CONDITIONS: Cigarette Smoking
Keywords: Ecological Momentary Assessment; mHealth; Smoking; Implementation Intentions
MeSH Terms: conditions — Cigarette Smoking; Smoking

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the Immediate Intervention, or Waitlist conditions. The Immediate Intervention participants receive the Ecological Momentary Intervention plus Implementation Intentions (EMI-II) immediately after randomization for two weeks, followed by two weeks of surveys. The Waitlist participants complete two weeks of surveys, followed by two weeks of receiving the EMAs plus EMI-II.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental): Participants in the Immediate Intervention condition will create their Implementation Intention (II) messages before the two-week EMA + EMI-II period begins. During the EMA + EMI-II period, participants will complete five daily EMAs, and they will also complete weekly assessments reporting their past week cigarette smoking as a distal outcome and rating intervention acceptability. Following the EMA + EMI-II period, participants will enter a two-week follow-up period. During this time, participants will not receive any messages, but will report past week smoking on a weekly basis.
  Interventions: Behavioral: Ecological Momentary Implementation Intentions Intervention (EMI-II)
- Waitlist (Active Comparator): Participants randomized to the Waitlist control condition will begin with a two-week no intervention condition during which they will report past week smoking on a weekly basis but will not receive any other intervention components. At the end of the two-week waitlist control period, participants will begin the two-week EMA plus EMI-II period. During the EMA plus EMI-II active study period, participants will complete five daily EMAs and weekly assessments to report their past week cigarette smoking and rate intervention acceptability. No follow-up is planned for the wait list control condition.
  Interventions: Behavioral: Ecological Momentary Implementation Intentions Intervention (EMI-II)

INTERVENTIONS:
Behavioral: Ecological Momentary Implementation Intentions Intervention (EMI-II) — To reduce smoking, this text messaging intervention will use a self-regulatory strategy, Implementation Intentions (II) to deliver appropriate alternative responses to cigarette smoking. Participants will create personalized II messages before starting the two-week intervention period. Then during the intervention period, after receiving Ecological Momentary Assessments (EMAs), participants will be micro-randomized to receive the EMI-II. During the EMA + EMI-II period, participants will complete five daily EMAs. After approximately 40% of these EMAs, participants will also receive the personalized EMI-II by text messaging.

SUMMARY:
This study will develop an ecological momentary implementation intentions intervention (EMI-II) for cigarette smoking, which will link critical situations where smoking is likely to occur with alternative responses to support avoidance of cigarette use. Using ecological momentary assessment (EMA) for data collection, this project will evaluate the feasibility, acceptability, and initial effectiveness of a micro-randomized trial (MRT) of EMI-II targeting cigarette smoking reduction in a sample of adults who smoke a minimum of 15 cigarettes per day (n=100).

DETAILED DESCRIPTION:
Cigarette smoking accounts for nearly 1 in 5 preventable deaths in the United States, and reducing cigarette smoking has been suggested for those not yet ready to quit. Cigarette reduction has been shown to longitudinally predict eventual cessation. Evidence suggests that smoking is highly sensitive to environmental stimuli, so ecological momentary interventions (EMI) embedded within daily life may help reduce cigarette smoking. Within the context of EMIs, researchers have explored different strategies to support smoking cessation and reduction. Implementation interventions (II) is a novel self-regulatory strategy that may help individuals reduce smoking. In II, individuals identify critical situations where smoking is likely to occur, then develop and plan appropriate alternative responses to avoid cigarette use. When II is delivered as a brief, single session intervention, II increases cessation rates relative to control conditions. Although II is well-suited for EMI because the brief messages are designed to be contextually relevant, no known research has evaluated whether repeated administration of II delivered by EMI reduces cigarette use. EMI-II may be beneficial with greater exposure and when delivered in the contexts where a behavior, such as smoking, is likely to occur.

This randomized controlled trial aims to test an ecological momentary implementation intentions intervention (EMI-II) to reduce cigarette smoking. This research seeks to identify in-the-moment intervention components that target momentary contextual and personal variables to effectively reduce cigarette smoking. Adults who smoke and are interested in reducing their cigarette use will be randomized to either the immediate intervention condition, or to a waitlist control. All participants will be followed for one month and will complete weekly surveys. Intervention participants will receive two weeks of the EMI-II with daily ecological momentary assessments (EMAs) in the two weeks post-randomization. Waitlist control participants will complete the weekly surveys for two weeks, then have access to the EMI-II with daily EMAs for two weeks. The daily EMAs are brief surveys in which participants report their current context and recent behavior and events.

This project consists of two primary aims:

Aim 1. To test the feasibility and acceptability of a customized, micro-randomized trial using EMI-II for smoking reduction.

The investigators hypothesize that at least 75% of participants who start the EMI-II component will complete the two-week active study period. Also, the investigators hypothesize that participants will rate the acceptability of the EMI-II at least a 3.5 out of 5, on average.

Aim 2. Test the initial effectiveness of EMI-II for reducing cigarette smoking.

The investigators hypothesize that participants receiving EMI-II will show greater reductions in self-reported smoking than participants assigned to an EMA-only control. In addition, the investigators hypothesize that self-reported cigarette smoking during the next EMA following EMI-II presentation will be lower, relative to cigarette smoking reported in EMAs that do not proximally follow the EMI-II delivery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English-language proficient
* Located in the United States
* Self-reports smoking 15 or more cigarettes per day in the past week
* Expresses interest in quitting or reducing smoking
* Has a cell phone with access to text messaging
* Willing to send and receive text messages related to smoking

Exclusion Criteria:

* Currently pregnant or plans to become pregnant
* Currently on psychotropic medications for smoking cessation
* Currently receiving behavioral treatment/therapy for smoking cessation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Saunders, PhD, Principal Investigator — Dartmouth College
Locations (1):
- Center for Technology and Behavioral Health, Dartmouth College, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Week 1 Follow-Up
Arm/Group | Immediate Intervention | Waitlist
Started | 39 | 41
Completed | 32 | 37
Not Completed | 7 | 4
Not completed — Lost to Follow-up | 7 | 4
Period: Week 2 Follow-Up
Arm/Group | Immediate Intervention | Waitlist
Started (If participants missed a follow-up, they were able to complete subsequent follow-ups.) | 39 | 41
Completed | 25 | 35
Not Completed | 14 | 6
Not completed — Lost to Follow-up | 14 | 6
Period: Week 3 Follow-Up
Arm/Group | Immediate Intervention | Waitlist
Started | 39 | 41
Completed | 23 | 30
Not Completed | 16 | 11
Not completed — Lost to Follow-up | 16 | 11
Period: Week 4 Follow-Up
Arm/Group | Immediate Intervention | Waitlist
Started | 39 | 41
Completed | 23 | 31
Not Completed | 16 | 10
Not completed — Lost to Follow-up | 16 | 10
Period: EMI-II Intervention
Arm/Group | Immediate Intervention | Waitlist
Started | 39 | 41
Completed | 25 | 31
Not Completed | 14 | 10
Not completed — Lost to Follow-up | 14 | 10

BASELINE CHARACTERISTICS:
Population: Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Intervention | Waitlist | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (1.5) | 40.0 (1.7) | 41.3 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 24 | 55
  Male | 8 | 17 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 37 | 38 | 75
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 5 | 5
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 33 | 33 | 66
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 41 | 80
Cigarettes smoker per day [Mean (Standard Deviation); unit: cigarettes smoked per day] | 30.2 (5.8) | 30.3 (7.2) | 30.2 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Completing Intervention Period
Description: To evaluate the feasibility of this customized EMI-II intervention, the investigators will examine the proportion of study participants completing the two-week intervention period, Week 2 in the Immediate Intervention arm and week 4 in the Waitlist arm.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Waitlist
Number analyzed (Participants) | 39 | 41
Participants | 25 | 31

2. Primary Outcome: Average Acceptability of the EMI-II Intervention
Description: To examine the acceptability of the EMI-II intervention, participants will rate the acceptability of the intervention on a Likert scale ranging from 1 (low acceptability) to 5 (high acceptability) on the two weekly surveys completed during the intervention period.
Time Frame: 2 weeks
Population: Includes participants who completed the AIM on the weekly surveys during the intervention period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Intervention | Waitlist
Number analyzed (Participants) | 24 | 28
score on a scale | 3.85 (0.84) | 3.55 (0.97)
Statistical Analysis 1: Comparison: Immediate Intervention vs Waitlist; Test type: Superiority; p = 0.24, t-test, 2 sided

3. Primary Outcome: Rate of Self-reported Cigarette Smoking
Description: Self-reported cigarette smoking will be assessed five times per day (morning, late morning, early afternoon, late afternoon, evening) during the intervention period. Participants will respond via text messaging to the question, "Since the last prompt, how many cigarettes have you smoked?"
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: cigarettes smoked per day
Arm/Group | Immediate Intervention | Waitlist
Number analyzed (Participants) | 22 | 28
cigarettes smoked per day | 30.3 (7.1) | 30.1 (5.0)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Immediate Intervention | Waitlist
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/41
Other Adverse Events (participants affected / at risk) | 0/39 | 0/41

LIMITATIONS AND CAVEATS:
More than twenty percent of participants were lost to follow-up before completing the final study survey.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT04967885/Prot_SAP_000.pdf